CLINICAL TRIAL: NCT05340998
Title: Radial accEss Crossover for PErcutaneous Coronary Procedures And ouTcome: the REPEAT Study
Acronym: REPEAT
Status: Completed | Type: Observational
Sponsor: Ospedale Sandro Pertini, Roma (Other)
Responsible Party: Principal Investigator, Alessandro Sciahbasi, MD, Principal Investigator, Ospedale Sandro Pertini, Roma
Other Study IDs: Pertini06
Record Dates: First submitted 2022-04-14; First posted 2022-04-22 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Coronary Angiography; Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Crossover Group: Patients with Transradial access failure for percutaneous coronary procedures necessitating vascular crossover
  Interventions: Procedure: Transradial access for percutaneous coronary procedures
- Non Crossover Group: Patients with successful transradial access for percutaneous coronary procedures
  Interventions: Procedure: Transradial access for percutaneous coronary procedures

INTERVENTIONS:
Procedure: Transradial access for percutaneous coronary procedures — Transradial approach for percutaneous coronary procedures. The modality of radial puncture (needle vs cannula), the choice of radial sheath (long vs short; hydrophilic vs non hydrophilic), the type of catheters employed, the use of spasmolytic agents and the choice of secondary vascular access will be left to the operator discretion

SUMMARY:
All patients who undergo to percutaneous coronary diagnostic or interventional procedures through transradial access (TRA) will be screened for inclusion in this prospective observational study and patients with TRA failure necessitating vascular crossover will be included in the Registry after signing a dedicated written informed consent. A Control group of consecutive patients with radial access and without crossover will be included. Primary end point of the study is the rate of in-hospital vascular complications and major bleeding in crossover vs non crossover groups

DETAILED DESCRIPTION:
All patients who undergo to percutaneous coronary diagnostic or interventional procedures through transradial approach (TRA) will be screened for inclusion in this prospective observational study and patients with TRA failure necessitating vascular crossover will be included in the Registry after signing a dedicated written informed consent. A Control group of consecutive patients with radial access and without crossover will be enrolled (2:1 rate compared to crossover group to avoid possible selection bias) after signing a dedicated written informed consent.

The modality of radial puncture (needle vs cannula), the choice of radial sheath (long vs short; hydrophilic vs non hydrophilic), the type of catheters employed, the use of spasmolytic agents and the choice of secondary vascular access will be left to the operator discretion.

According to the selected secondary access, patients will be divided in two groups: patients with a secondary (or tertiary) wrist access (total wrist Group) and patients with a crossover to femoral (Femoral Group). Patients included in the total wrist group may have a secondary access to the ulnar artery (ipsilateral or contralateral) or to the contralateral radial.

All patients will be checked during the procedure, immediately after and 24 hour post to evaluate possible vascular complications and bleeding.

Patient baseline characteristics, hospital data, comorbid conditions and complications will be recorded in a dedicated electronic case report form.

Exclusion criteria will be: lack of signed informed consent, age <18 years.

Primary End point of the study is the rate of in-hospital vascular complications and major bleeding in crossover vs non crossover groups.

Secondary End-points are:

* The rate of vascular complications or bleeding in total wrist vs femoral Group.
* The rate of minor bleeding
* Procedure duration
* Fluoroscopy time
* Number of catheters employed
* Differences among operators and Centers

Vascular complications are defined as any vascular damage clinically documented as vessel perforation, arterial-venous fistula, pseudoaneurysm, arterial dissection, retroperitoneal hematoma and compartmental syndrome. Major bleeding complications are defined according to the BARC classification, as BARC 3 (overt bleeding plus a hemoglobin drop > 3 g/dL; any transfusion with overt bleeding, cardiac tamponade; bleeding requiring surgical intervention for control; bleeding requiring intravenous vasoactive agents and intracranial haemorrhage) and BARC 5 (fatal bleeding).

Minor bleeding is defined as Hematoma larger than 10 cm not requiring medical intervention (Easy III)

ELIGIBILITY:
Inclusion Criteria:

* All patients who undergo to percutaneous coronary diagnostic or interventional procedures through transradial access

Exclusion Criteria:

* Lack of signed informed consent, age <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an indication to percutaneous coronary procedures performed through transradial approach
Sampling Method: Non-Probability Sample
Enrollment: 1357 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-16 (Actual)

PRIMARY OUTCOMES:
Vascular complications and major bleeding | up to seven days
  The rate of in-hospital vascular complications and major bleeding in crossover vs non crossover groups

SECONDARY OUTCOMES:
Minor bleeding | up to seven days
  The rate of minor bleeding in crossover vs non crossover groups

CONTACTS AND LOCATIONS:
Locations (10):
- Italy (10):
  - Ospedale di Avezzano, Avezzano
  - Ospedale S. Andrea, Roma
  - Ospedale S. Camillo, Roma
  - Ospedale Sandro Pertini, Roma
  - Ospedale Santo Spirito, Roma
  - Policlinico Agostino Gemelli, Roma
  - Policlinico Umberto I, Roma
  - Ospedale di Sassari, Sassari
  - Ospedale di Teramo, Teramo
  - Ospedale di Trento, Trento